CLINICAL TRIAL: NCT01738776
Title: Nutritional Risk Factors for Hip Fracture: a Case Control Study
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Anne Torbergsen, Clinical Nutritionist, Oslo University Hospital
Other Study IDs: S-0916901(REK); 120000MM (Other Grant/Funding Number: Oslo University Hospital)
Record Dates: First submitted 2012-11-14; First posted 2012-11-30 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Hip Fracture
Keywords: hip fracture; risk factors; vitamin K1; vitamin D; bone turnover markers; osteocalcin; undercarboxylated osteocalcin; bone specific alkaline phosphatase (BALP); insulin like growth factor 1 (IGF1); parathyroid hormone (PTH)
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — For vitamin and hormone analysis serum was collected For some vitamin analysis EDTA blood was collected For RNA analysis fullblood was collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Hip fracture patients participating in a randomised controlled trial (RCT) of orthogeriatric care (ClinicalTrials.gov NCT01009268)
- Controls: A group of voluntary elderly persons without a history of hip fracture, recruited specifically for this purpose

SUMMARY:
Low Body Mass Index (BMI) is a risk factor for hip fracture, but it is unknown if it is the low BMI per se that increases risk of hip fracture or if specific micro-nutrients contribute. The investigators want to elucidate this aspect in a case control study studying micronutrients in serum and bone turnover markers of hip fracture patients compared with controls of the same age.

ELIGIBILITY:
Inclusion Criteria:

Cases are admitted acutely for a femoral neck fracture, a trochanteric or a subtrochanteric femoral fracture.

Exclusion Criteria:

* Hip fracture as part of multi-trauma or high energy trauma (defined as a fall from a higher level than 1 metre). One recent fracture in addition to the hip fracture (e.g. radius or shoulder) is acceptable.
* Regarded as moribund at admittance.
* Absence of a valid informed consent or assent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cases: The first 116 patients of an ongoing RCT were included consecutively and examined by blood samples pre operatively for nutrition and hormone analysis. The catchment area for the cases was the city of Oslo, Norway.
  A control group, at the same age with no history of hip fracture, was drawn at random from inhabitants aged 60 - 100 years (median age 82 years) at the census files of Oslo in 2005.
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
micronutrient association with increased risk of hip fracture | At admission
  Blood was drawn for micronutrient analysis in hip fracture patients and in controls

SECONDARY OUTCOMES:
Are micronutrients related to bone turnover markers | At admission
  Blood was drawn for bone turnover analysis. Correlation analysis with micronutrients was performed

CONTACTS AND LOCATIONS:
Overall Officials: Morten Mowe, PhD, Study Chair — Oslo University Hospital
Locations (1):
- University of Oslo, Institute of Clinical Medicine, Oslo, Norway

REFERENCES:
- [Derived] Torbergsen AC, Watne LO, Frihagen F, Wyller TB, Mowe M. Effects of nutritional intervention upon bone turnover in elderly hip fracture patients. Randomized controlled trial. Clin Nutr ESPEN. 2019 Feb;29:52-58. doi: 10.1016/j.clnesp.2017.11.012. Epub 2018 Oct 30. PMID 30661701
- [Derived] Torbergsen AC, Watne LO, Wyller TB, Frihagen F, Stromsoe K, Bohmer T, Mowe M. Micronutrients and the risk of hip fracture: Case-control study. Clin Nutr. 2017 Apr;36(2):438-443. doi: 10.1016/j.clnu.2015.12.014. Epub 2015 Dec 23. PMID 26795217